CLINICAL TRIAL: NCT03630601
Title: A Pilot Study of Photoacoustic Imaging (PAI)
Brief Title: Photoacoustic Imaging in Diagnosing Changes in Tumors in Participants With Breast Cancer, Sarcoma, Skin Cancer, or Soft Tissue Malignancy and Healthy Volunteers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Diagnostic issues
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I 56617; NCI-2018-01424 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 56617 (Other: Roswell Park Cancer Institute); R01CA204636 (NIH)
Record Dates: First submitted 2018-07-24; First posted 2018-08-15 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Breast Carcinoma; Healthy Subject; Malignant Soft Tissue Neoplasm; Sarcoma; Skin Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (photoacoustic imaging) (Experimental): Participants undergo PAI on different parts of the body over 20 minutes for up to 5 imaging sessions for 6 months.
  Interventions: Procedure: Photoacoustic Imaging

INTERVENTIONS:
Procedure: Photoacoustic Imaging — Undergo PAI

SUMMARY:
This pilot trial studies how well photoacoustic imaging works in diagnosing changes in tumors in participants with breast cancer, sarcoma, skin cancer, or soft tissue malignancy and healthy volunteers. Photoacoustic imaging is a low-risk imaging method that provides information about the oxygenation of tissues using a combination of light and ultrasound techniques. Photoacoustic imaging uses a signal from hemoglobin to provide information on blood flow and oxygen levels, and it may be helpful in determining changes in tumors after chemotherapy or radiation treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the feasibility of the current photoacoustic imaging (PAI) technology in various groups of human subjects.

SECONDARY OBJECTIVES:

I. To define the utility of the current PAI on various groups of human subjects.

II. When possible, via means of an existing data review, PAI will be correlated with standard imaging modalities performed on patients as routine part of clinical care or on protocol.

III. When possible, via means of an existing data review, PAI will be compared to pathologic specimens.

IV. When possible, via means of an existing data review, PAI data will be correlated with outcomes of patients to therapies they receive.

OUTLINE:

Participants undergo PAI on different parts of the body over 20 minutes for up to 5 imaging sessions for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* ALL GROUPS:
* No restriction on race or ethnic background.
* Subject must understand the investigational nature of the study and sign an independent Ethics Committee/Institutional Review Board approved written informed consent prior to receiving any study related procedure.
* HEALTHY VOLUNTEERS:
* No history of antimicrobial therapy or drug treatment including anti-hypertensive, diuretic, immunosuppressive or anti-depressant drugs in the previous 6-month period.
* No history of diabetes.
* No history of cancer to the body site to be imaged.
* BREAST, SARCOMA, SKIN CANCER, AND SUPERFICIAL MALIGNANCY PATIENTS:
* Biopsy-proven aforementioned malignancy.
* SURGICAL FLAP PATIENTS:
* Need for plastic surgery reconstruction with a free or rotational flap.

Exclusion Criteria:

* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Unwilling or unable to follow protocol requirements or provide consent.
* Any condition which in the Investigator's opinion deems the subject an unsuitable candidate to undergo imaging procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of photoacoustic imaging (PAI) to quantify tumor characteristics | Up to 6 months
  This will be deemed a success if at least 3 imaging sessions produce a usable image. Usable datasets will be defined as those images with detectable PAI signal with minimal or no artifacts within the region of interest. This analysis will be done in the imaged sample, consisting of enrolled patients who attempt at least one imaging session. Patients who do not attempt at least one imaging session will be replaced.

SECONDARY OUTCOMES:
Utility of serial PAI measurements | Up to 6 months
  This will be explored by comparison with disease and outcome characteristics collected during routine cancer treatment, including standard imaging modalities, pathology results, and clinical outcomes. Results of these analyses are intended to inform development of early stage (Phase 1/2) clinical trials that consider PAI summaries as biomarkers for treatment response.
Serial PAI oxygenation measurements | Up to 6 months
  This will be correlated with disease and patient characteristics using Analysis of Variance (ANOVA ) for categorical factors
Serial PAI oxygenation measurements | Up to 6 months
  This will be correlated with disease and patient characteristics using OLS regression for continuous factors
Serial PAI oxygenation measurements | Up to 6 months
  This will be correlated with disease and patient characteristics using Cox Regression models for progression and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States